CLINICAL TRIAL: NCT07312591
Title: Using Line@ Online Platform to Follow up on Counseling Intervention Effectiveness for Illegal Drug Use Among College and University Students
Brief Title: Using the LINE@ Online Platform to Follow Up on Illegal Drug Use Among College and University Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Principal Investigator, Li Yi Xuan, Principal Investigator, National Taiwan Normal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 202506HM023
Record Dates: First submitted 2025-09-16; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Illegal Drug Use

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LINE@ Online Platform Intervention Group (Experimental): LINE@ Online Platform Intervention
  Interventions: Device: LINE@ Online Platform Intervention
- Control Group (No Intervention)

INTERVENTIONS:
Device: LINE@ Online Platform Intervention — Using digital learning materials covering family functioning, substance dependence severity, motivation for change, and emotional health management.
  Arms: LINE@ Online Platform Intervention Group

SUMMARY:
This study developed a LINE@ online platform for tracking college and university students involved in illegal drug use, with the aim of evaluating the effectiveness of the intervention.

DETAILED DESCRIPTION:
Effectiveness indicators were collected using a structured questionnaire, including family functioning, severity of substance dependence, motivation for change, and emotional health management. In addition, a structured questionnaire was used to gather university students' user evaluations of the LINE@ online platform.

ELIGIBILITY:
Inclusion Criteria:

* College students with a history of illegal drug use (confirmed by urine screening or other methods, such as self-reported use, curiosity-driven misuse, or accidental use)

Exclusion Criteria:

* Younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Family Functioning | To be completed within 2 months from the start of participation
  1.Assessment of family dynamics and functioning using using validated scales FAMILY APGAR (questionnaire). 2.The score ranges from 0 to 10, with higher scores indicating better family functioning.
Severity of Substance Dependence | To be completed within 2 months from the start of participation
  1.Evaluation of the severity of substance dependence among participants using validated scales The Severity of Dependence Scale (questionnaire). 2.The score ranges from 0 to 15, with higher scores indicating a greater level of substance dependence in the participant.
Motivation for Change | To be completed within 2 months from the start of participation
  1.Measurement of participants' motivation to change their substance use using validated scales University of Rhode Island Change Assessment (questionnaire). 2.The score ranges from 2 to 10, with higher scores indicating a greater severity of addictive behaviors and a higher level of motivation to change in the participant's clinical course.
Emotional Health Management | To be completed within 2 months from the start of participation
  1.Assessment of emotional health management skills through using validated scales Brief Symptom Rating Scale (questionnaire). 2.The score ranges from 0 to 20, with higher scores indicating a greater level of emotional distress.
Drug Abuse Screening Test | To be completed within 2 months from the start of participation
  1.Survey on illegal drug use in the past 1 month using validated scales Drug Abuse Screening Test (questionnaire). 2.The score ranges from 0 to 10, with higher scores indicating a higher risk level of illegal drug use.

SECONDARY OUTCOMES:
User Evaluation of the LINE@ Online Platform | To be completed within 2 months from the start of participation
  1.Participants' evaluation of the usability and effectiveness of the LINE@ platform using validated scales System usability scale (questionnaire). 2.The score ranges from 0 to 100, with higher scores indicating a higher evaluation of the educational material by the participants.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Normal University, Taipei, Heping E. Rd, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided